CLINICAL TRIAL: NCT04766684
Title: A Randomized, Comparison Study of L.M.X.4 Cream Versus J-Tip Needle-Free Injection System With Lidocaine in Children Undergoing In-Office Percutaneous Achilles Tenotomy for Clubfoot
Brief Title: Comparison Study of LMX4 Cream Versus J-Tip Needle-Free Injection System With Lidocaine for In-Office PAT for Clubfoot
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Martus, Associate Professor of Orthopaedic Surgery and Rehabilitation, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200842
Record Dates: First submitted 2021-01-26; First posted 2021-02-23 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Clubfoot
Keywords: Clubfoot; J-Tip
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: On the day of or after the final casting visit, the participant will be randomized in equal proportion (1:1) to either the control group (receive L.M.X.4 cream with J-Tip saline injection) or the intervention group (placebo cream with J-Tip with 0.25mL of 1% Xylocaine MPF). Researchers, physicians, nurses, CCLS, caregivers, and patients will be blinded to which group the patient is assigned to. The only person who will remain unblinded is the research coordinator.
  An outside pharmacy, the Health & Wellness Compounding Pharmacy, will provide and blind the L.M.X.4 and placebo creams. The Vanderbilt Investigational Drug Service will provide the blinded J-Tip 1% Xylocaine MPF and saline vials. The Investigational Drug Service will store the creams provided by the outside pharmacy and the J-Tip vials. They will assist in dispensing the creams/vials to the outpatient clinic.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- J-Tip with 0.25mL of 1% Xylocaine MPF with placebo cream (Experimental)
  Interventions: Device: J-Tip with Xylocaine MPF with placebo cream
- L.M.X.4 cream with J-Tip saline injection (Active Comparator)
  Interventions: Drug: L.M.X.4 cream with J-Tip saline injection

INTERVENTIONS:
Device: J-Tip with Xylocaine MPF with placebo cream — J-Tip with 0.25mL of 1% Xylocaine MPF with placebo cream
  Arms: J-Tip with 0.25mL of 1% Xylocaine MPF with placebo cream
Drug: L.M.X.4 cream with J-Tip saline injection — L.M.X.4 cream with J-Tip saline injection
  Arms: L.M.X.4 cream with J-Tip saline injection

SUMMARY:
Infants undergoing Ponseti treatment for idiopathic clubfoot often require percutaneous tendoachilles lengthening (TAL) after serial casting. This procedure is commonly performed in the office with a local anesthetic to avoid exposure to general anesthesia in the operating room. Topical anesthetic creams are commonly used to provide local analgesia for this procedure. The cream is applied to the infant's skin around the heel cord and requires 30-60 minutes to provide adequate analgesia, reaching a depth of up to 5 mm at maximum effect. Alternative to analgesic cream, the J-tip is a needle-free jet injection system that uses compressed CO2 instead of a needle to push 0.25 ml of lidocaine into the skin, providing local analgesia at the site of administration. This method likewise provides analgesia to the site of application at a depth of 5-8 mm, yet only takes approximately 1-2 minutes to achieve maximum effect.

Aim 1: Determine which pain management method, L.M.X.4 Cream vs. J-tip 1% Xylocaine MPF Injection, provides the greatest pain relief to infants with clubfoot undergoing an in-office percutaneous TAL. Hypothesis: J-tip 1% Xylocaine MPF injection will provide equal or greater pain control when compared to L.M.X.4 cream in infants undergoing an in-office percutaneous TAL.

Aim 2: Determine if there is a difference in the rate of adverse events between the two pain management methods, L.M.X.4 Cream vs. J-tip 1% Xylocaine MPF Injection.

Hypothesis: J-tip 1% Xylocaine MPF injection will not be associated with an increased rate of adverse events in comparison to L.M.X.4 cream in infants undergoing an in-office percutaneous TAL.

If J-tip Xylocaine MPF injection is shown to provide comparable or better pain control without an increase in adverse events, use of this needle-free injection system will decrease the overall length of visit and the cost of the procedure, thus increasing the quality, safety, and value.

DETAILED DESCRIPTION:
Clubfoot is a common congenital birth deformity, with a prevalence of 1 in 1000 live births. If left untreated, clubfoot can cause significant disability. Treatment of clubfoot has evolved over several decades and now favors the method of serial casting pioneered by Ignacio Ponseti. This technique involves weekly stretching followed by application of a long leg cast. In the majority of cases, percutaneous tendoachilles lengthening (TAL) is required to correct the equinus component of the clubfoot deformity. Following TAL, a long leg cast is applied for 3 weeks and then a foot-abduction orthosis is utilized to maintain correction of the deformity.

Percutaneous TAL can be performed in the operating room under general anesthesia or in an outpatient setting utilizing local or topical anesthesia. While studies have shown that in-office percutaneous TAL is safe and efficient, little has been done to investigate the pain management strategies implemented for infants during this procedure. Pain management for infants during procedures is important because it has been shown that repeated painful exposures during early stages of life can lead to alterations in hemodynamic stability, altered stress hormone expression, heightened peripheral sensitivity, altered pain reactivity that persists following the painful stimulus, and somatization. One study identified the infant's ability to become conditioned to painful stimuli, such as heel sticks, at as early as 3 days old. Based on this, providers should be prepared to provide adequate pain management for infants during painful procedures, such as in-office TAL, by utilizing non-pharmaceutical techniques, pharmaceutical techniques, or a combination of both.

Needle injection of local anesthetic is generally avoided prior to an in-office percutaneous TAL due to the needle puncture and the concern that soft tissue swelling may prevent accurate palpation of the heel cord during the procedure. As such, topical local anesthetic creams are commonly used to provide local analgesia for this procedure. The cream is applied to the infant's skin around the heel cord and requires 30-60 minutes to provide adequate analgesia, reaching a depth of up to 5 mm at maximum effect. At our institution, a 5 gram tube of L.M.X.4 cream costs $4.12, while other studies report that a larger 25 gram tube of EMLA cream can cost as much as $56, with the excess being wasted. Alternative to anesthetic cream, the J-tip is a needle-free jet injection system that uses compressed CO2 instead of a needle to push 0.25 ml of lidocaine into the skin, providing local analgesia at the site of administration. This method provides analgesia to the site of application at a depth of 5-8 mm and takes approximately 5 minutes to achieve maximum effect. At our institution, the cost of the J-tip applicator and a 20 mL 1% lidocaine vial is $5.11. Multiple studies have demonstrated the J-Tip to provide greater pain control than other pharmaceutical options, including EMLA cream and vapocoolant ("freezy") spray.

The goal of this study is to determine if the J-Tip Xylocaine MPF injection provides equal or greater pain control in clubfoot patients undergoing an in-office percutaneous TAL when compared to L.M.X.4 cream, without an increase in adverse events. If this is true, use of J-tip Xylocaine MPF injection will decrease the overall time and cost of the visit, while ultimately increasing the quality, safety, and value of in-office TAL for the treatment of clubfoot in infants.

ELIGIBILITY:
Inclusion Criteria

* Clubfoot patients less than 6 weeks of age at start of casting
* Patients presenting to Vanderbilt DOT 4 Clinic for care
* Patients undergoing in-clinic Achilles Tenotomy

Exclusion Criteria

* Clubfoot patients greater than 6 weeks of age at the start of casting
* Previous clubfoot treatment
* Patients with a neuromuscular condition (spina bifida, caudal regression syndrome, arthrogryposis, etc.)
* In-office TAL is not recommended by treating physician due to patient factors such as age or size

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
FLACC (Face, Legs, Activity, Cry, Consolability) Scale | Baseline, before cast placement to tenotomy procedure at the end of casting, approximately 10 weeks.
  The FLACC scale is used to assess pain in children. For this study, it will be administered by the Certified Child Life Specialist. The Face, Legs, Activity, Cry, Consolability (FLACC) scale is a measurement used to assess pain in children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. Lower values represent lessening pain on the scale
Pulse Oximetry | Baseline, before cast placement to tenotomy procedure at the end of casting, approximately 10 weeks.
  Pulse oximetry will be used to measure oxygen levels in the blood. An oxygen saturation level of 95 percent is considered normal

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Martus, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Children's Orthopaedics, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan to share IPD with other researchers.

REFERENCES:
- [Background] Taddio A, Shah V, Gilbert-MacLeod C, Katz J. Conditioning and hyperalgesia in newborns exposed to repeated heel lances. JAMA. 2002 Aug 21;288(7):857-61. doi: 10.1001/jama.288.7.857. PMID 12186603
- [Background] Spanos S, Booth R, Koenig H, Sikes K, Gracely E, Kim IK. Jet Injection of 1% buffered lidocaine versus topical ELA-Max for anesthesia before peripheral intravenous catheterization in children: a randomized controlled trial. Pediatr Emerg Care. 2008 Aug;24(8):511-5. doi: 10.1097/PEC.0b013e31816a8d5b. PMID 18645542
- [Background] COMMITTEE ON FETUS AND NEWBORN and SECTION ON ANESTHESIOLOGY AND PAIN MEDICINE. Prevention and Management of Procedural Pain in the Neonate: An Update. Pediatrics. 2016 Feb;137(2):e20154271. doi: 10.1542/peds.2015-4271. Epub 2016 Jan 25. PMID 26810788
- [Background] Morcuende JA, Dolan LA, Dietz FR, Ponseti IV. Radical reduction in the rate of extensive corrective surgery for clubfoot using the Ponseti method. Pediatrics. 2004 Feb;113(2):376-80. doi: 10.1542/peds.113.2.376. PMID 14754952
- [Background] Lunoe MM, Drendel AL, Levas MN, Weisman SJ, Dasgupta M, Hoffmann RG, Brousseau DC. A Randomized Clinical Trial of Jet-Injected Lidocaine to Reduce Venipuncture Pain for Young Children. Ann Emerg Med. 2015 Nov;66(5):466-74. doi: 10.1016/j.annemergmed.2015.04.003. Epub 2015 Apr 29. PMID 25935844
- [Background] Lebel E, Karasik M, Bernstein-Weyel M, Mishukov Y, Peyser A. Achilles tenotomy as an office procedure: safety and efficacy as part of the Ponseti serial casting protocol for clubfoot. J Pediatr Orthop. 2012 Jun;32(4):412-5. doi: 10.1097/BPO.0b013e31825611a6. PMID 22584844
- [Background] Herzenberg JE, Radler C, Bor N. Ponseti versus traditional methods of casting for idiopathic clubfoot. J Pediatr Orthop. 2002 Jul-Aug;22(4):517-21. PMID 12131451
- [Background] Ansar A, Rahman AE, Romero L, Haider MR, Rahman MM, Moinuddin M, Siddique MAB, Mamun MA, Mazumder T, Pirani SP, Mathias RG, Arifeen SE, Hoque DME. Systematic review and meta-analysis of global birth prevalence of clubfoot: a study protocol. BMJ Open. 2018 Mar 6;8(3):e019246. doi: 10.1136/bmjopen-2017-019246. PMID 29511012

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT04766684/Prot_SAP_002.pdf
  • Informed Consent Form (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04766684/ICF_003.pdf